CLINICAL TRIAL: NCT03665571
Title: Ex Vivo Expansion of Natural Killer Cells From Blood in Patients With Pancreatic Cancer and the Evaluation of Killing Activity of Expanded Natural Killer Cells
Brief Title: Evaluation of Killing Activity of Expanded Natural Killer Cells From Blood in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Professor, Asan Medical Center
Other Study IDs: 2015-0865
Record Dates: First submitted 2018-09-03; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Natural killer cell and plasma from peripheral blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Activation method: NK cell was incubated with either K562 cells
  Interventions: Diagnostic Test: Receptor specific activation method
- Receptor specific activation method: NK cell was incubated with P815-ULBP1+CD48 cells that trigger NK cell synergy via NKG2D and 2B4
  Interventions: Diagnostic Test: Receptor specific activation method

INTERVENTIONS:
Diagnostic Test: Receptor specific activation method — NK cell was incubated with P815-ULBP1+CD48 cells that trigger NK cell synergy via NKG2D and 2B4

SUMMARY:
Pancreatic cancer, one of the deadliest epithelial malignancies, has a 5-year survival rate of only about 8%. The mortality rate has decreased slightly, but the incidence rate has been steadily increasing, and it is predicted to be the second leading cause of cancer mortality in 2030. Early diagnosis of pancreatic cancer and the development of innovative therapies are needed, and various basic and clinical studies based on pancreatic cancer biology are underway. Recently, studies on the effect of natural killer (NK) cells on cancer progression and the development of therapeutic agents using them have been actively conducted. NK cells are a component of innate lymphoid cells, accounting for approximately 5-15% of total peripheral blood mononuclear cells (PBMC).

DETAILED DESCRIPTION:
Investigators will apply a new method to evaluate the activity of NK cells in pancreatic cancer patients, and to analyze the correlation with the progression of the tumor and the prognosis of the patient. And investigators will analyze the multifactorial factors affecting the activity of NK cells and conducted this study to help establish new diagnostic and therapeutic strategies for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient who is admitted to the pancreatic surgery department for the treatment of pancreas tumor
* Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.
* Life expectancy of at least 6 months based on discretion of treating
* Adequate hematologic function defined by the following laboratory parameters: Hemoglobin > 100, Platelet count > 100 and Absolute granulocyte count > 1.5.

Exclusion Criteria:

* Patients who received preoperative chemotherapy or radiotherapy.
* Previous or concurrent malignancies.
* Any serious medical condition within 6 months prior to study entry such as myocardial infarction, uncontrolled congestive heart failure, unstable angina, serous infection.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pancreatic ductal adenocarcinoma Mucinous adenocarcinoma Neuroendocrine carcinoma Adenosquamous carcinoma Mucinous cystic neoplasm Intraductal mucinous neoplasm Solid pseudopapillary neoplasm Neuroendocrine tumor Serous cystic neoplasm Benign cyst Chronic pancreatitis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
NK cell activity | 1 month before operation
  In order to compare the activity of NK cells according to the activation method, NK cells obtained from the blood of participants will be analyzed. Investigates will use two methods to analysis the activity of NK cell by FACS (Fluorescence-activated cell sorting). The degree of expression of CD107a on the cell surface and the degree of IFN-γ secretion will be compared by FACS.

SECONDARY OUTCOMES:
Tumor recurrence | two year after tumor diagnosis
  In order to analyze the correlation of NK cell activity with the prognosis of the participants, investigators will follow up the recurrence of the tumor. This will be analyzed with the activity of NK cell.
Survival of participants | two year after tumor diagnosis
  In order to analyze the correlation of NK cell activity with the prognosis of the participants, investigators will follow up the survival of the patients. This will be analyzed with the activity of NK cell.

CONTACTS AND LOCATIONS:
Overall Officials: Song Cheol Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided